CLINICAL TRIAL: NCT01919554
Title: Investigation of the Safety and Tolerability of Sublingual Immunotherapy Tablets of House Dust Mite Allergen Extracts in Adolescents With House Dust Mite-associated Allergic Rhinitis
Brief Title: Safety Study of Sublingual Immunotherapy Tablets of House Dust Mite Allergen Extracts in Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stallergenes Greer (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VO73.13
Record Dates: First submitted 2013-08-02; First posted 2013-08-09 (Estimated); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2015-12

CONDITIONS: Allergic Rhinitis Due to House Dust Mite
Keywords: House Dust Mite Allergic Rhinitis; Phase I; House Dust Mite Allergen Extract
MeSH Terms: interventions — Sublingual Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 500 IR (Experimental): 500 IR house dust mites allergen extract tablet
  Interventions: Biological: 500 IR house dust mites allergen extract tablet
- 1000 IR (Experimental): 1000 IR house dust mites allergen extract tablet
  Interventions: Biological: 1000 IR house dust mites allergen extract tablet
- 1500 IR (Experimental): 1500 IR house dust mites allergen extract tablet
  Interventions: Biological: 1500 IR house dust mites allergen extract tablet
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Biological: Placebo tablet

INTERVENTIONS:
Biological: 500 IR house dust mites allergen extract tablet — One sublingual tablet daily during 10 days
  Other Names: Sublingual immunotherapy tablet
  Arms: 500 IR
Biological: 1000 IR house dust mites allergen extract tablet — Two sublingual tablets daily during 10 days
  Other Names: Sublingual immunotherapy tablet
  Arms: 1000 IR
Biological: 1500 IR house dust mites allergen extract tablet — Three sublingual tablets daily during 10 days
  Other Names: Sublingual immunotherapy tablet
  Arms: 1500 IR
Biological: Placebo tablet — One, two or three sublingual placebo tablets daily during 10 days matching with the sublingual immunotherapy tablets
  Other Names: Sublingual placebo tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of different doses of sublingual tablets of house dust mite (HDM) allergen extracts in adolescents with house dust mite-associated allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from patient and parent(s)/legal representative.
* Male or female patient from 12 to 17 years.
* Diagnosed rhinitis with medical history consistent with HDM-induced allergic rhinitis for at least 1 year before visit 1
* Positive Skin Prick Test to House Dust Mites(HDM)and HDM-specific IgE serum value ≥ 0.7 kUnit/L.
* Concommittant controlled asthma allowed up to GINA 1 or 2 treatment step
* Spirometry with best FEV1 > 80% of predicted FEV1.

Exclusion Criteria:

* Patient with a nasal or oral disease that could interfere with the safety assessments
* Patient has undergone recent nasal surgery
* Patient with asthma receiving therapy consistent with GINA (Global INitiative for Asthama) treatment step 3, 4, or 5.
* Patient with partially controlled or uncontrolled asthma
* Patient with a past or current disease, which as judged by the Investigator, may affect the patient's participation in or the outcome of this study.
* Female patient pregnant or breast-feeding/lactating.
* Female patient of childbearing potential planning a pregnancy during this trial or not using a medically accepted contraceptive method.
* Patient treated with beta-blockers, tricyclic antidepressants or monoamine oxidase inhibitors (MAOIs).
* Patient who received allergy specific immunotherapy for house dust mites for more than 1 month in the 5 years before screening or who is currently receiving immunotherapy with any allergen.
* patient with a history of anaphylaxis
* patient having participated in any clinical study within the 12 weeks before visit 1

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Piyush Patel, MD, Principal Investigator — Inflamax Research Incorporated
Locations (1):
- Inflamax Research Inc., Mississauga, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient First Visit 29 JUL 2013, Last Patient Last Visit 30 SEP 2013
Period: Overall Study
Arm/Group | 500 IR | 1000 IR | 1500 IR | Placebo
Started | 9 | 9 | 9 | 10
Completed | 9 | 9 | 8 | 9
Not Completed | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Set: All patients who received at least one dose of treatment including those who did not complete the study were included in the Safety Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | 500 IR | 1000 IR | 1500 IR | Placebo | Total
Number analyzed (Participants) | 9 | 9 | 9 | 10 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.4 (1.33) | 14.1 (1.45) | 15.3 (1.12) | 14.6 (1.78) | 14.9 (1.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 5 | 7 | 19
  Male | 6 | 5 | 4 | 3 | 18

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability Evaluated on Treatment Emergent Adverse Events
Description: Safety and tolerability evaluated on the number of participants who reported at least one treatment-emergent adverse event (TEAE)
Time Frame: 10 dosing treatment days
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | 500 IR | 1000 IR | 1500 IR | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 10
participants | 4 | 6 | 9 | 4

2. Secondary Outcome: Treatment Emergent Serious Adverse Events
Description: Treatment emergent Serious Adverse Events
Time Frame: 10 dosing treatment days
Measure: Number; unit: participants
Arm/Group | 500 IR | 1000 IR | 1500 IR | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 10
participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Adverse Events Leading to Study Withdrawal
Description: Incidence of adverse events leading to study withdrawal
Time Frame: 10 dosing treatment days
Measure: Number; unit: participants
Arm/Group | 500 IR | 1000 IR | 1500 IR | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 10
participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | 500 IR | 1000 IR | 1500 IR | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 4/9 | 6/9 | 9/9 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 500 IR (N=9) | 1000 IR (N=9) | 1500 IR (N=9) | Placebo (N=10)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 5 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Oral pruritus (Gastrointestinal disorders) | 1 | 4 | 3 | 0
Lip pruritus (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Oedema mouth (Gastrointestinal disorders) | 2 | 1 | 2 | 0
Lip oedema (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Tongue eruption (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 2 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Ear pruritus (Ear and labyrinth disorders) | 2 | 1 | 2 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 2 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 2
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No